CLINICAL TRIAL: NCT05423704
Title: DAHANCA Proton Feasibility Study
Brief Title: Feasibility of Patient Selection and Treatment of Head-neck Cancer With Proton Therapy in Denmark
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA proton feasibility
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Head-and-neck Cancer
Keywords: Proton radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiotherapy (Experimental): Proton radiotherapy according to the guidelines defined by the Danish Head-Neck Cancer Group (DAHANCA). Treatment: 66-68 Gy/ 33-34 fx/ 6/W,with cisplatin 40 mg/m2/W and nimorazole to suitable patients
  Interventions: Other: Proton radiotherapy

INTERVENTIONS:
Other: Proton radiotherapy — Proton radiotherapy according to the guidelines defined by the Danish Head-Neck Cancer Group (DAHANCA). Treatment: 66-68 Gy/ 33-34 fx/ 6/W, with cisplatin 40 mg/m2/W and nimorazole to suitable patients

SUMMARY:
A study to investigate feasibility of local selection of patients with squamous cell carcinoma of the pharynx or larynx using anticipated benefit of proton radiotherapy in reducing the risk of late dysphagia or xerostomia.

DETAILED DESCRIPTION:
In preparation for a randomised study in Denmark (DAHANCA 35) the feasibility of selecting newly diagnosed patients with squamous cell carcinoma of the pharynx or larynx for proton therapy at the local treatment centers is investigated. A proton and a photon doseplan is prepared for patients planned for primary radiotherapy . If proton radiotherapy reduces the anticipated absolute risk of dysphagia >= grade 2 (DAHANCA scale and/or xerostomia >= grade 2 (EORTC Head-Neck 35) with a clinical relevant value the patient is offered proton therapy at the Danish Center for Particle Therapy. The anticipated risk of xerostomia and dysphagia is estimated using Normal-Tissue Complication Models (NTCP).

At least five patients from each of the six Danish centers are required in this feasibility study.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically proven squamous cell carcinoma of the pharynx or larynx planned for primary radiotherapy with curative intent

A predicted clinical significant reduction in the risk of any of the two primary endpoints (>= grade 2 observer-rated dysphagia or grade 2 patient-reported xerostomia) after proton therapy compared to photon therapy based on comparison of the individual patient dose plans

No current or earlier malignancies, which may influence treatment, evaluation or outcome of the head-neck cancer

Informed consent as required by law

Above 18 years of age

Exclusion Criteria:

Patient with cancers of the glottic larynx (stage I/II), skull base, sino-nasal area, nasopharynx, unknown primary tumor and prior malignancies.

Patients with contraindications for proton therapy (as per 2019 pacemakers, implanted defibrillators and tracheostomy)

Inability to attend full course of radiotherapy or follow-up visits in the outpatient clinic

Distant metastasis

Previous radiotherapy of the head and neck

Previous surgery for the primary cancer with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Dysphagia >= grade 2 | Six months after end of radiotherapy
  The rate of observer-reported dysphagia >= grade 2 measured by the DAHANCA late toxicity score (grade 0-4, with 0 being best)
Xerostomia = grade 2 | Six months after end of radiotherapy
  The rate of patient-reported xerostomia measured by the EORTC Quality of life questionnaire (QLQ) Head-Neck (HN) 35 (grade 1-4, with 1 being best)

SECONDARY OUTCOMES:
Loco-regional tumor control | Up to five years after end of radiotherapy
  Time to event of local-regional failure, from date of randomization to the date of first documented loco-regional failure.
  Rates are estimated by the Kaplan-Meier method. Interim analyses after 100, 200 and 300 patients. Will not be reported before the primary endpoint.
Overall survival | Up to five years after end of radiotherapy]
  From date of randomisation to date of death
Acute toxicity | From the beginning of and up to two months after end of radiotherapy]
  DAHANCA acute toxicity score (grade 0-4, 0 being best)
Late toxicity | From two months to five years after end of radiotherapy]
  DAHANCA late toxicity score (grade 0-4, 0 being best)
EORTC QLQ-Head-Neck 35 | Up to five years after end of radiotherapy
  Swallowing and social-eating scale and specific HN35 items related to eating and pain (grade 1-4, 1 being best)
EORTC C30 | Up to five years after end of radiotherapy]
  Specific C30 items related to fatigue, nausea and vomiting (grade 1-4, 1 being best)
Time from referral to treatment | From date of referral to proton treatment to first proton treatment (Assessed up to 60 days)
  Time from referral to proton center to first proton treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Friborg, MD, PhD, Principal Investigator — Danish Head-Neck Cancer Group (DAHANCA)
Locations (7):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Danish Center for Particle Therapy, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Næstved Hospital, Næstved
  - Odense University Hospital, Odense